CLINICAL TRIAL: NCT00388375
Title: Can Ultrasound be Used as an Alternative to Chest Radiography After Central Venous Catheter Insertion to Confirm Proper Catheter Position and to Exclude Pneumothorax?
Brief Title: Can Ultrasound be Used to Verify CVC Position and to Exclude Pneumothorax?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not feasible, did not have the study population.
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25185
Record Dates: First submitted 2006-10-12; First posted 2006-10-16 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2012-11

CONDITIONS: Catheterization, Central Venous
MeSH Terms: interventions — High-Energy Shock Waves

ARMS (1):
- CVC Internal Jugular or Subclavian Vein (No Intervention)
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — limited ultrasound examination to evaluate the following areas: Examination of the subclavian and internal jugular veins to assess proper catheter placement PTX detection, using lung sliding and comet-tail artifact Visualization of the heart (right atrium and ventricle) and the inferior vena cava through the subcostal window

SUMMARY:
The purpose of this study is to determine if emergency room physicians can use bedside ultrasound to quickly determine the proper placement of a central venous catheter and to evaluate for complications such as a punctured lung.

DETAILED DESCRIPTION:
Central venous catheterization (CVC) of the subclavian or internal jugular veins is a common procedure performed in the emergency department (ED). This procedure is followed by complications in 0.3 to 12% of cases. Pneumothorax (PTX) and catheter-tip misplacement can occur. The diagnosis of these complications requires a chest radiograph (CXR). In certain cases, CXR may be time-consuming, requiring more than 30 minutes. This could be harmful in the case of critically ill patients. Moreover, several investigators have questioned the need of routine post-procedural CXR in the absence of clinical complications.

Recent data has shown that ultrasound can accurately detect PTX in critically ill patients. Furthermore, bedside ultrasound is an easy technique to investigate the subclavian and internal jugular veins, and can improve the success rate of catheter insertion. Ultrasound also allows visualization of central venous catheters in vivo. Ultrasound has been reported as a tool to detect catheterization complications and misplacement when performed by ICU physicians, but has never been studied in the ED.

This method could be valuable in hemodynamically unstable patients, who quickly need a CVC for the measurement of central venous pressure, immediate fluid resuscitation, and infusion of vasoactive medications. Similarly, bedside ultrasound examination could quickly confirm PTX and allow immediate chest tube insertion in case of respiratory distress after catheter insertion.

We hypothesize that bedside ultrasound examination performed by ED physicians could accurately detect placement of the CVC and the presence or absence of a PTX after catheterization of the jugular and subclavian veins.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older
* Signed consent
* In need of subclavian or internal jugular central line placement

Exclusion Criteria:

* Any subject who refuses or whose family refuses to sign consent
* Any subject in whose immediate transfer from the care of the ED to another location is mandated by clinical presentation
* Any subject under the age of 18
* Any subject being evaluated for chest trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The presence or absence of a misplaced CVC as detected by US and CXR. | 10 Minutes
The presence or absence of PTX as detected by US and CXR | 10 minutes

SECONDARY OUTCOMES:
Time needed to complete the US exam and CXR | varies

CONTACTS AND LOCATIONS:
Overall Officials: Jason Nomura, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Heath System, Newark, Delaware, United States